CLINICAL TRIAL: NCT03953443
Title: INST 1008: Expression and Epigenetic Silencing of MicroRNA for Predicting the Therapeutic Response and Prognosis of HPV-negative Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Expression & Epigenetic Silencing of MicroRNA for Predicting Therapeutic Response and Prognosis of HPV-negative HNSCC
Status: Completed | Type: Observational
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST 1008
Record Dates: First submitted 2019-05-08; First posted 2019-05-16 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh HNSCC tumor-distant normal mucosal tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not interventional

SUMMARY:
A two-part molecular epidemiological study will be conducted to comprehensively assess the association between miR expression and miR promoter methylation and the response to therapy and prognosis in primary, HPV-negative HNSCC patients. Part 1 will be a prospective collection of 25 pairs of fresh tumor-distant normal mucosal tissue in patients with HNSCC. Ultimately, 15 HPV-negative tumor-mucosal pairs will be utilized for discovery work in identifying miRs whose expression is up- or down-regulated in tumors. Part 2 will test the association between miR expression and miR promoter methylation, and therapeutic response and survival in all archived surgical cases of HPV-negative HNSCC at University of New Mexico Hospital (UNMH) collected after 1990.

DETAILED DESCRIPTION:
* Part 1, Prospective Collection of Fresh Tumor-Distant Normal Pairs

The investigators will prospectively collect 25 pairs of fresh HNSCC tumor-distant normal mucosal tissue.

* Part 2, Retrospective Molecular Epidemiology Study of the Association of miRs with Therapeutic Response and Prognosis in HNSCC.

The investigators will comprehensively test the association between miR expression and miR promoter methylation, and the response to therapy and survival in all cases of surgical HPV-negative HNSCC at UNMH collected after 1990. Lip and nonkeratinizing nasopharyngeal cases will be excluded as these are etiologically distinct and related to cutaneous SCC or to EB virus infection, respectively. No cases will be excluded due to gender, age, race or ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a known or suspected diagnosis of HNSCC

  * Any primary site may be included, except nonkeratinizing nasopharyngeal SCC or lip SCC.
  * Patients are planned for diagnostic biopsies for suspected HNSCC, or for therapeutic surgery for HNSCC.
  * Patients are naïve to radiation to the head and neck, prior to research biopsies.
  * Patients have not received chemotherapy for the diagnosis of HNSCC, prior to research biopsies.
* Age > 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Patients sign an informed consent, agreeing to fresh tumor biopsy as well as distant normal mucosal biopsy for purposes of described research. Research biopsies will be in addition to planned surgery. In cases where tumor resection is planned, a representative part of the tumor will be submitted for research purposes.

Exclusion Criteria:

* Nonkeratinizing nasopharyngeal carcinoma
* Lip squamous cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected HNSCC
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2010-12-17 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Identify tumor specific microRNAs (miRs) whose expression increases or decreases by over 2 fold in fresh tumor vs. distant normal mucosa from patients with head and neck squamous cell carcinoma (HNSCC) negative for human papillomavirus (HPV) | As long as needed to collect 15 HPV-negative tumor-mucosal sample pairs and complete sequencing, up to 10 years
  SOLiD sequencing of fresh tumor-distant normal pairs will discover miRs whose expression is altered in HNSCC tumors. SOLiD sequencing will provide fully quantitative data for the expression of known and novel miRs. Because HPV-related tumors comprise approximately 20% of all HNSCC and are biologically distinct from HPV negative tumors classically associated with tobacco and alcohol, only HNSCC without p16 overexpression will be used in this discovery experiment. This restriction will increase homogeneity of the samples and the power to detect miRs associated with the etiology of HPV-negative HNSCC. The miRs identified will be validated using qPCR assay in the tumor-normal pairs and in p16-negative HNSCC cell lines (n>15). In addition, miRs previously reported to be dysregulated in HNSCC will be subjected to similar validation, even if not identified during the SOLiD sequencing discovery phase.
Identify miRs whose reduced expression in HPV-negative HNSCC is due to promoter methylation | As long as needed to complete sequencing and analyze results, up to 5 years
  miRs with reduced expression in tumor tissue identified under Outcome 1 will be scrutinized for CpG rich promoters by checking the UCSC database. The methylation status of CpG rich promoters of miRs will be examined by COBRA assay in tumor vs. normal pairs (n=15) and in p16-negative HNSCC cell lines (n>15). The heterogeneity of methylation status across the CpG rich promoter will be characterized by bisulfate sequencing using the COBRA PCR product. The silencing of miRs by promoter methylation will be examined by comparing mean miR expression levels between the methylation categories for the tumor-normal pairs and for the HNSCC cell lines. This is primarily a descriptive study.
Define the statistical association between the expression of tumor specific miRs, miR methylation, and the therapeutic response and prognosis of HPV-negative HNSCC using patient medical records | As long as needed to collect and analyze information from medical records, up to 5 years
  The therapeutic response and prognosis of HPV-negative HNSCC will be collected from two sources: the patient's case file from the New Mexico Tumor Registry (NMTR) and from the patient's UNMH medical record. qRT PCR will be designed to quantify the miR expression in RNA extracted from the formalin-fixed, paraffin embedded (FFPE) tissues. A methylation-specific PCR (MSP) will be designed to facilitate the large-scale methyl-typing in all retrospective clinical samples. The primary analysis will be performed in HPV-negative HNSCC. A secondary analysis will be conducted to include all HNSCC, with and without p16 overexpression. p16 overexpression status will be adjusted in the secondary analysis. The association between miR expression status (high or low) and miR methylation status (yes or no), and patient's PFS and OS will be examined using Kaplan-Meier survival plots and the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Garth Olson, MD, Principal Investigator — University of New Mexico Comprehensive Cancer Center
Locations (1):
- University of New Mexico - Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No